CLINICAL TRIAL: NCT02569086
Title: Population Pharmacokinetics of Piperacillin in the Early Phase of Severe Sepsis - Does Standard Dosing Result in Therapeutic Plasma Concentrations?
Brief Title: Piperacillin PK Analysis in Severe Sepsis Patients
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Kristina Öbrink-Hansen, MD, University of Aarhus
Other Study IDs: PIP/TAZO-INTERMEDIATE
Record Dates: First submitted 2015-09-30; First posted 2015-10-06 (Estimated); Results first posted 2017-11-13 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2015-10

CONDITIONS: Sepsis; Severe Sepsis
Keywords: Sepsis; Therapeutic Drug Monitoring; Beta-lactams; Pharmacokinetics
MeSH Terms: conditions — Sepsis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Blood draw

SUMMARY:
Antibiotic dosing in septic patients poses a challenge for clinicians due to the pharmacokinetic changes seen in this population. Piperacillin/tazobactam is often used for empirical treatment, and initial appropriate dosing is crucial for reducing mortality.

The investigators aim was to determined the pharmacokinetic profile of piperacillin 4g every 8 hour in 22 patients treated empirically for sepsis and severe sepsis. A PK population model was be established with the dual purpose to assess current standard treatment and to simulate alternative dosing regimens and modes of administration. Time above the minimal inhibitory concentration (T>MIC) predicted for each patient was evaluated against clinical breakpoint MIC for Pseudomonas Aeruginosa (16 mg/L). Pharmacokinetic-pharmacodynamic (PK-PD) targets evaluated were 100% f T>MIC and 50% fT>MIC.

DETAILED DESCRIPTION:
Appropriate empiric antibiotic therapy is crucial for reducing mortality in septic patients. Pathophysiological changes associated with the septic process, i.e. changes in volume of distribution (Vd), protein binding and drug clearance (Cl), lead to pharmacokinetic (PK) alterations that may influence the efficacy of the drug. As a consequence, antibiotic plasma concentrations are variable and hard to predict in this patient population. Optimal dosing and exposure can therefore be a challenge and standard antibiotic dosing regimens may result in subtherapeutic concentrations and therapeutic failure. Appropriate dosing is also essential in order to maximize bacterial killing and minimize development of antimicrobial resistance.

Piperacillin/tazobactam is a β-lactam-β-lactamase inhibitor combination with extended-spectrum antibacterial activity, which is often used for empirical treatment of severe infections. The antibacterial activity is time-depentent, i.e. the activity is related to the time for which the free unbound drug concentration is maintained above the minimum inhibitory concentration (MIC) (fT>MIC). By maximizing T>MIC, therapeutic impact increases and the risk of drug resistance development is reduced (7). For β-lactams, a fT>MIC of at least 50% is associated with clinical efficacy. However, higher targets may be needed for maximal bactericidal effect in critically ill patients. Piperacillin/tazobactam is by standard practice administered as intermittent bolus infusion (IB). However, prolonged infusion, both extended infusion (IE) and continuous infusion (CI) is believed to optimize drug exposure and has a PK advantage compared to IB.

Patients with known or suspected sepsis or severe sepsis, treated empirically with piperacillin/tazobactam 4g/0,5g (Tazocin®) every eight hour (q8h) were eligible for the study. Piperacillin/tazobactam (4g/0,5g) was administered intravenously (i.v.) as a 3-minute bolus infusion . Serial blood samples were collected over one dosing interval for up to three consecutive days if piperacillin/tazobactam treatment was maintained.

The free concentrations of piperacillin in sera were assessed using ultra high performance liquid chromatography (UHPLC).

Clinical MIC breakpoints according to the European Committee on Antimicrobial Susceptibility Testing (EUCAST) for Pseudomonas aeruginosa were used to evaluate the following PK/PD targets: 100% f T>MIC and 50% fT>MIC.

There was no intervention in the study.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with Piperacillin/Tazobactam 4g/0.5g every 8 hour for less than 48 hours

Exclusion Criteria:

* renal replacement therapy
* Age under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe sepsis treated empirically with Piperacillin/Tazobactam
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merete Storgaars, MD, PhD, Study Director — Department of Infectious Diseases, Aarhus University Hospital, Denmark
Locations (1):
- Department of Infectious Diseases, Aarhus University Hospital, Denmark, Aarhus, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andersen MG, Thorsted A, Storgaard M, Kristoffersson AN, Friberg LE, Obrink-Hansen K. Population Pharmacokinetics of Piperacillin in Sepsis Patients: Should Alternative Dosing Strategies Be Considered? Antimicrob Agents Chemother. 2018 Apr 26;62(5):e02306-17. doi: 10.1128/AAC.02306-17. Print 2018 May. PMID 29507062

RESULTS

PARTICIPANT FLOW:
Groups:
- Piperacillin Pharmacokinetics: Patients with known or suspected sepsis or severe sepsis, treated empirically with piperacillin/tazobactam 4g/0,5g (Tazocin®) every eight hour (q8h).
Period: Overall Study
Arm/Group | Piperacillin Pharmacokinetics
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Piperacillin Pharmacokinetics
Number analyzed (Participants) | 22
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [33 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 12
Body weight [Median (Inter-Quartile Range); unit: kg] | 76 [64 to 82]
estimated creatinine clearance (eCLCr) [Median (Inter-Quartile Range); unit: mL/minute] | 106 [46 to 152]

OUTCOME MEASURES:

1. Primary Outcome: 100% f T>MIC: Free Piperacillin Concentration Maintained Above the MIC Throughout the Dosing Interval.
Description: The piperacillin plasma concentration-time profiles were best described by a two-compartment model. Each individual model predicted T>MIC was compared to clinical breakpoint MIC for P.aeruginosa (16 mg/L). The number of patients who achieved the pre-defined PK/PD target were reported.
Time Frame: Participants will be followed to day five (120 hours) after initiation of piperacillin/tazobactam treatment.
Measure: Number; unit: participants
Arm/Group | Piperacillin Pharmacokinetics
Number analyzed (Participants) | 22
participants | 4

2. Primary Outcome: 50% f T>MIC: Free Piperacillin Concentration Maintained at a Level Four Times Above the MIC 50% of the Dosing Interval.
Description: as for outcome 1
Time Frame: Participants will be followed to day five (120 hours) after initiation of piperacillin/tazobactam treatment.
Measure: Number; unit: participants
Arm/Group | Piperacillin Pharmacokinetics
Number analyzed (Participants) | 22
participants | 15

ADVERSE EVENTS:
Arm/Group | Piperacillin Pharmacokinetics
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes